CLINICAL TRIAL: NCT05626634
Title: A Phase 2, Multicenter, Open-label, Long-term Safety Study of LP352 in Subjects With Developmental and Epileptic Encephalopathy Who Completed Study LP352-201 and Are Candidates for Continuous Treatment for Up to 52 Weeks
Brief Title: Open-label, Long-term Safety Study of LP352 in Subjects With Developmental and Epileptic Encephalopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Longboard Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP352-202
Record Dates: First submitted 2022-11-15; First posted 2022-11-25 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Developmental and Epileptic Encephalopathy; Dravet Syndrome; Lennox-Gastaut Syndrome
Keywords: CDKL5 deficiency disorder; developmental and epileptic encephalopathy; Dravet Syndrome; epilepsy; Lennox-Gastaut Syndrome; treatment resistant epilepsy; tuberous sclerosis complex
MeSH Terms: conditions — Epilepsies, Myoclonic; Lennox Gastaut Syndrome; CDKL5 deficiency disorder; Epilepsy; Tuberous Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LP352, bexicaserin (Experimental): Subjects will be titrated up to highest tolerated dose of LP352 during a 15-day period, followed by a 48-week maintenance period and a 15-day taper/down titration period.
  Interventions: Drug: LP352, bexicaserin

INTERVENTIONS:
Drug: LP352, bexicaserin — LP352 6 mg, 9 mg or 12 mg administered three times daily, orally or through G-tube

SUMMARY:
The objective of this study is to assess the long-term safety, tolerability, and efficacy of adjunctive therapy of LP352 in subjects with developmental and epileptic encephalopathies who completed participation in Study LP352-201.

DETAILED DESCRIPTION:
This Phase 2, multicenter, open-label, multiple-dose extension clinical study is designed to evaluate long-term safety of LP352 in subjects with developmental and epileptic encephalopathy who completed Study LP352-201.

The study consists of a Screening Period (Day -1) and a 50-week open-label Treatment Period that includes a 15-day Up-titration Period (during which time subjects will titrate up to their highest tolerated doses) and an open-label Maintenance Period (48 weeks). The Treatment Period will be followed by a Down-titration/Taper Period (up to 15 days) and Follow-up Period (14 days after completion of down-titration). The starting dose of up-titration will be 6 mg TID. The target final maintenance doses are 6 mg TID, 9 mg TID, and 12 mg TID after a 15-day up-titration period, if tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female, age 12 to 65 years who have satisfactorily completed study LP352-201
2. Diagnosis of Dravet syndrome, Lennox-Gastaut syndrome, or other developmental and epileptic encephalopathy
3. The patient/parent/caregiver is able and willing to attend study visits, complete the diary and take study drug as instructed

Exclusion Criteria:

1. Had an SAE in Study LP352-201 that was definitely, probably, or possibly related to exposure to study drug
2. Current or past history of cardiovascular or cerebrovascular disease, such as cardiac valvulopathy, myocardial infarction, stroke, pulmonary arterial hypertension or abnormal blood pressure
3. Has glaucoma, renal impairment, liver disease or any other medical condition that would affect study participation or pose a risk to the subject
4. Current or recent history of moderate or severe depression, anorexia nervosa, bulimia or at risk of suicidal behavior
5. Currently taking anorectic agents, monoamine oxidase inhibitors; serotonin agonists or antagonists including fenfluramine, atomoxetine, vortioxetine, or other medications for weight loss
6. Positive test result on the drug screen, except tetrahydrocannabinol (THC) for patients taking prescribed cannabidiol

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent Adverse Events | Baseline up to Week 52
  Incidence and severity of treatment-emergent adverse events, including serious adverse events and adverse events leading to study discontinuation and clinically significant changes in vital signs, physical examination endpoints, clinical safety laboratory values and ECGs
Columbia-Suicide Severity Rating Scale (C-SSRS) Response | Baseline up to Week 52
  Type of Suicidal Ideation, Intensity (1 - 5, with 5 being most severe), Suicidal Behavior
Patient Health Questionnaire-9 Total Score and Question 9 Score | Baseline up to Week 52
  Severity Rating Scale: 0 - 27; higher scores indicate greater severity of depressive disorder

SECONDARY OUTCOMES:
Percent Change from Baseline in Observed Countable Motor Seizure Frequency During the Treatment Period | Baseline to Week 50
  Baseline Used for Seizure Frequency = Baseline from Study LP352-201 and Baseline from Study LP352-202
Proportion of Subjects with > 50% Reduction in Total Seizures During the Treatment Period | Baseline to Week 50
Percent Reduction in Individual Seizure Type During the Treatment Period | Baseline to Week 50
Proportion of Subjects Requiring Rescue Medication During the Treatment Period | Baseline to Week 50
Percent Change from Baseline in the Number of Episodes of Status Epilepticus During the Treatment Period | Baseline to Week 50
Percent of Subjects with Countable Motor Seizure-free Days During the Treatment Period | Baseline to Week 50
Percentage Change from Baseline in Non-motor and Difficult to Count Seizures | Baseline to Week 50
LGS: Percentage Change from Baseline in the Frequency of Observed Drop Seizures Over the Treatment Period | Baseline to Week 50

CONTACTS AND LOCATIONS:
Overall Officials: Dennis J Dlugos, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (28):
- United States (25):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Rancho Los Amigos National Rehabilitation Center (RLANRC), Downey, California
  - University of California San Francisco, San Francisco, California
  - Northwest Florida Clinical Research Group, Gulf Breeze, Florida
  - University of Miami, Miami, Florida
  - Advent Health Orlando, Orlando, Florida
  - Research Institute of Orlando, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Spectrum Health, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Boston Children's Health Physicians LLP, Hawthorne, New York
  - Northwell Health, New York, New York
  - Northeast Regional Epilepsy Group, Staten Island, New York
  - OnSite Clinical Solutions LLC, Charlotte, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Providence Neurological Specialties-East, Portland, Oregon
  - Child Neurology Consultants of Austin, Austin, Texas
  - Austin Epilepsy Care Center, Austin, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Washington Valley Medical Center, Renton, Washington
- Australia (3):
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Austin Health, Heidelberg, Victoria
  - Alfred Health, Melbourne, Victoria